CLINICAL TRIAL: NCT04955275
Title: The Efficacy of a Remote Cognitive Remediation Therapy (CRT) Program on Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BHS-1660
Record Dates: First submitted 2021-06-17; First posted 2021-07-08 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease Patients receiving Cognitive Remediation Therapy (Experimental): Parkinson's Disease Subjects will undergo 10 weeks of Brain HQ training, 2 times a week an hour at a time. Also patients pre- and post-intervention RBANS and PDQ-39 scores.
  Interventions: Other: Cognitive Remediation Therapy Program (BrainHQ)
- Parkinson's Disease Patients not receiving Cognitive Remediation Therapy (No Intervention): Parkinson's Disease Subjects will receive no intervention, but still undergo pre- and post-intervention RBANS and PDQ-39 scores.

INTERVENTIONS:
Other: Cognitive Remediation Therapy Program (BrainHQ) — Brain HQ games involving training cognitive abilities like memory and attention, made up of adapting tasks or creating our own.
  Arms: Parkinson's Disease Patients receiving Cognitive Remediation Therapy

SUMMARY:
Purpose/Goal: To determine if a remote computerized cognitive remediation program (CRT) can stabilize or improve cognitive functioning in a group of patients from the New York Institute of Technology Academic Health Care Center with Parkinson's disease (PD) after three months of intervention.

Hypothesis: Patients with PD who present with current cognitive deficits will show improvement in such deficits after three months of participation in a remotely supervised structured Cognitive Remediation Therapy Program (CRT) compared to control subjects with PD who receive treatment as usual.

Research design: Pilot study. Prospective randomized treatment and control comparison pre-post study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be currently enrolled in the Rock Steady Boxing Program at the Adele Smithers Parkinson's Disease Center.
2. Subjects must be between 40 and 85 years old (including both ages) at the time of study screening.
3. Subjects must have a diagnosis of Parkinson's disease by a physician.
4. Subjects must have a MOCA score of 20 or above.
5. Subjects must demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in this research study.
6. Subjects must have been clinically stable for 2 weeks prior to consent; in the judgment of the Investigator.
7. Subjects must have the visual, auditory, and motor capacity to use the intervention in the judgment of the Principal Investigator.
8. Subjects must be technologically capable of utilizing a computer and navigating through the programs.
9. Subjects must be mechanically capable of utilizing a computer and computer mouse.

Exclusion Criteria:

1. Subjects should not be participating in a concurrent research study or other interventional clinical trial 30 days prior to consenting.
2. Subjects should not have a history of mental retardation or pervasive developmental disorder; or other co-morbid neurological disorder (e.g., epilepsy.)
3. Subject is unable to physically use a computer or a computer mouse.
4. Subject is unable to or refuses to give consent.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Pre-Intervention | Initially, before any intervention/start of study.
  A brief, individually administered test measuring attention, language, visuospatial/constructional abilities, and immediate and delayed memory.
The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Post-Intervention | 10 weeks after intervention/completion of the study.
  A brief, individually administered test measuring attention, language, visuospatial/constructional abilities, and immediate and delayed memory.
Parkinson's Disease Questionnaire (PDQ-39) Pre-Intervention | Initially, before any intervention/start of study.
  A test that assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication.
Parkinson's Disease Questionnaire (PDQ-39) Post-Intervention | 10 weeks after intervention/completion of the study.
  A test that assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication.
Montreal Cognitive Assessment (MOCA) Pre-Intervention Screening | Initially, before any intervention/start of study.
  A rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diez-Cirarda M, Ibarretxe-Bilbao N, Pena J, Ojeda N. Efficacy of cognitive rehabilitation in Parkinson's disease. Neural Regen Res. 2018 Feb;13(2):226-227. doi: 10.4103/1673-5374.226390. No abstract available. PMID 29557365
- [Background] Diez-Cirarda M, Ojeda N, Pena J, Cabrera-Zubizarreta A, Lucas-Jimenez O, Gomez-Esteban JC, Gomez-Beldarrain MA, Ibarretxe-Bilbao N. Increased brain connectivity and activation after cognitive rehabilitation in Parkinson's disease: a randomized controlled trial. Brain Imaging Behav. 2017 Dec;11(6):1640-1651. doi: 10.1007/s11682-016-9639-x. PMID 27757820
- [Background] Petersen RC, Caracciolo B, Brayne C, Gauthier S, Jelic V, Fratiglioni L. Mild cognitive impairment: a concept in evolution. J Intern Med. 2014 Mar;275(3):214-28. doi: 10.1111/joim.12190. PMID 24605806
- [Background] Gough N, Brkan L, Subramaniam P, Chiuccariello L, De Petrillo A, Mulsant BH, Bowie CR, Rajji TK. Feasibility of remotely supervised transcranial direct current stimulation and cognitive remediation: A systematic review. PLoS One. 2020 Feb 24;15(2):e0223029. doi: 10.1371/journal.pone.0223029. eCollection 2020. PMID 32092069
- [Background] Milman U, Atias H, Weiss A, Mirelman A, Hausdorff JM. Can cognitive remediation improve mobility in patients with Parkinson's disease? Findings from a 12 week pilot study. J Parkinsons Dis. 2014;4(1):37-44. doi: 10.3233/JPD-130321. PMID 24322063

DOCUMENTS (1):
  • Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04955275/ICF_000.pdf